CLINICAL TRIAL: NCT05536219
Title: Impact of the Presence of Anti-interferon Autoantibodies on the Viral Load in Severe Respiratory Infections in Intensive Care
Brief Title: Impact of the Presence of Anti-interferon Autoantibodies on the Viral Load in Severe Respiratory Infections
Acronym: INTERFERICUS
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0674
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Severe Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Nasopharyngeal swab
  * Venous blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Serum anti-IFN-I antibodies — Anti-IFN-I autoantibodies presence will be assessed through serological methods (ThermoFisher Kit)

SUMMARY:
Type I interferons (IFN-I) production is induced by the detection of viral molecules, such as RNA or DNA viral strands, through pattern recognition receptors (PRR) present on many immune cell types. Despite a minimal concentration, IFN-I secretion activate the secretion, by neighbouring cells, of more than 700 proteins with antiviral properties (inhibition of viral replication, destabilization of virus membranes, etc.). IFN-I constitute therefore one of the major first line of defence established by the immune system in response to viral infection. Briefly, during the Coronavirus disease (COVID-19) pandemic, several teams including ours, highlighted a lack of IFN-I response in approximately one in five individuals presenting a severe form of COVID-19.

Interestingly, within a large part of them, in vitro investigations revealed the presence of autoantibodies presenting neutralizing capacities against alpha and/or omega interferons This finding confirms the deleterious role of anti-IFN-I autoantibodies on the antiviral immune response and the key role of IFN-I pathway regarding defences against COVID-19 infection. Furthermore, those observations pave the way to interesting research that would allow understanding the underlying pathophysiological mechanisms of severe viral respiratory infection.

The research hypothesis are:

i) IFN-I deficiency could induce severe forms of viral infections which could lead to intensive care admission ii) IFN-I deficiency could increase viral loads in nasopharyngeal samples, and be associated with protracted viral clearance iii) The frequency of viral co-infections may be higher in case of IFN-I antiviral pathway blockade, iv) severe forms of respiratory viruses' infections could be induced by other anti-cytokine autoantibodies.

In addition to confirming research hypotheses recently mentioned, the aim of this clinical protocol will be to assess the impact of antiviral innate immune response alterations in severe respiratory infections.

ELIGIBILITY:
Inclusion Criteria:

For adult patients :

* Patients with acute respiratory failure requiring the administration of oxygen* to maintain peripheral oxygen saturation at at least 90%

  * in patients with chronic respiratory failure, an oxygen flow higher than the usual flow or a duration of non-invasive ventilation longer than the usual duration will be required.
* Patients with influenza, RSV or SARS-CoV-2 infection diagnosed by Reverse Transcription Polymerase Chain Reaction (RT-PCR) or antigen test in the last 7 days
* Patients hospitalized in participating intensive care units

For pediatric patient :

* In respiratory distress placed on oxygen with signs suggestive of viral infection:

  1. moderate or absent fever or nasopharyngeal congestion or cough
  2. signs of acute respiratory distress (polypnea > 2DS of the normal value, intercostal drawing, thoraco-abdominal sway) with more or less marked hypoxia (SpO2 < 92% under ambient air),
  3. and/or significant apnea (associated with bradycardia or desaturation),
  4. and/or dietary difficulties (reduction of rations to less than 50% of the usual ration).
* Hospitalized in the pediatric emergency and intensive care unit of Hôpital Femme Mère Enfant (HFME)

Exclusion Criteria:

* Opposition of the patient or his close family/friend to inclusion in the study

  * Patient under legal protection measure
  * Patient who was included in this study during a previous stay
  * Immunodepression defined by: bone marrow allograft less than 24 months old, chemotherapy for less than 6 months, HIV infection with CD4<200/mm3 or <15%, corticosteroid therapy for more than 2 weeks with a daily dose greater than 10 mg of prednisolone equivalent, immunosuppressive treatment administered in the previous 3 months (6 months for rituximab), aplasia, asplenia or splenectomy.
  * Patient under 30 kg (for adults) and less than 3 kg (for children)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients and pediatric patients admitted to intensive care unit with acute respiratory failure induced by RSV, influenza or SARS-Cov-2 viral infection (for adults only) or in respiratory distress placed on oxygen with suggestive sign(s) of viral infection for minors only.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-08-08 (Estimated); Study Completion 2027-08-08 (Estimated)

PRIMARY OUTCOMES:
Change in viral load in nasopharyngeal samples for adult patients | At Day 0 and Day 7
  Main outcome will be the difference of viral load (expressed in log copies per million cells) at D0±1 day and D7±1 day post inclusion (presence or absence of anti-IFN-I autoantibodies), and stratified by pathogen (influenza, respiratory syncytial virus (RSV), COVID-19).
Change in viral load in nasopharyngeal samples for pediatric patients | At Day 0 and Day 7
  Main outcome will be the prevalence of anti-interferon antibodies presence (expressed in log copies per million cells) at Day 0 and Day 7 post inclusion and to compare the respiratory co-infections frequency.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Femme Mère et enfant, Bron, Rhone
  - Hopital Lyon Sud, Pierre-Bénite, Rhone
  - Hôpital Croix Rousse, Lyon, Rhône